CLINICAL TRIAL: NCT06547983
Title: Effectiviteit en Beleving Van FooDIYou
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TNO (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #2023-083
Record Dates: First submitted 2024-08-02; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: Digital studies; Personalized nutrition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- Intervention group (Experimental)
  Interventions: Other: Personalized nutritional advice
- Intervention plus group (Experimental)
  Interventions: Other: Personalized nutritional advice and food boxes

INTERVENTIONS:
Other: Personalized nutritional advice — Participants in the intervention group received personalized nutrition advice based on their dietary habits, weight, anthropometric data and physical activity.
  Arms: Intervention group
Other: Personalized nutritional advice and food boxes — Participants in the intervention plus group received the personalized nutrition advice while also receiving food boxes which are composed based on the personalized nutritional advice.
  Arms: Intervention plus group

SUMMARY:
Studies have shown that personalized nutrition advice is more effective compared to generic nutrition advice for weight loss purposes. However, since decentralization of clinical trials is on the rise, it of interest to test whether personalized nutrition advice is as effective when provided fully digitally. In the current study the investigators compare the effects of generic vs. personal nutritional interventions in a fully digital study. Three groups are included, a control group receiving generic nutritional advice, an intervention group receiving personalized nutrition advice and an intervention plus group receiving personalized nutrition advice plus personalized meals. The trial takes six weeks. Anthropometric data are collected every two weeks and data on changes in nutritional diet are collected at the beginning and end of the intervention. In addition, the opinion of the participants on trial participation is asked as well every two weeks during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-60 years
* BMI between 25 and 40
* Motivated to lose weight
* Can fill in a digital questionnaire
* Posses a smartphone, computer, weighing scale and measuring tape to perform anthropometric measurements.

Exclusion Criteria:

* Any food allergy
* Chronic diseases influencing food intake (e.g., IBD)
* Participating in another intervention study
* Females in menopausal transition
* Follow a specific diet

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Body weight in kilograms | 6 weeks

SECONDARY OUTCOMES:
Body height in meters | 6 weeks
BMI as calculated by combining body weight and height (kg/m^2) | 6 weeks
Hip circumference in centimeters | 6 weeks
Waist circumference in centimeters | 6 weeks
Neck circumference in centimeters | 6 weeks
Wrist circumference in centimeters | 6 weeks
Dietary habits as measured using the Nutri+ Module | 6 weeks
  Nutri+ Module is a food frequency questionnaire developed by TNO (TNO, Leiden, The Netherlands). This is used to obtain information on the habitual total food intake by asking food category consumption over the day.
Opinion on digital intervention as measured using an online questionnaire. | 6 weeks
  The online questionnaire contained the following questions and multiple choice answers:
  * How easily can the participant implement the nutritional advice? (very easily/easily/moderately/poorly/very poorly)
  * How pleasant is it to implement the nutritional advice? (very pleasant, pleasant, moderate, unpleasant, very unpleasant)
  * Did participant's diet change compared to before the intervention? (Yes/no)
  * Does the participant feel like the participant's diet is healthier compared to before the intervention? (Yes/no)
  * How easily can the participant perform the anthropometric measurements by themselves? (very easily/easily/moderately/poorly/very poorly)
  * Are the questions in the questionnaire clear? (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Femke Hoevenaars, PhD, Principal Investigator — TNO
Locations (1):
- TNO, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Jong JC, Hoevenaars FP, Peters LG, Berendsen CM, Pasman WJ, Caspers MP, Dulos R, Wopereis S. A Real-Life Digital Intervention for Personalized Nutrition in Adults With Overweight or Obesity: Remote Randomized Controlled Trial. J Med Internet Res. 2026 Jan 5;28:e73367. doi: 10.2196/73367. PMID 41490780